CLINICAL TRIAL: NCT02727998
Title: Combining Neurobiology and New Learning: Ketamine and Prolonged Exposure: A Potential Rapid Treatment for Post Traumatic Stress Disorder (PTSD)
Brief Title: Intensive 7-day Treatment for PTSD Combining Ketamine With Exposure Therapy
Acronym: PTSD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study ran out of funding
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1509016530; 23260 (Other Grant/Funding Number: NARSAD)
Record Dates: First submitted 2016-03-14; First posted 2016-04-05 (Estimated); Results first posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Single infusion of Ketamine with prolonged exposure (Experimental): After the reactivation of the scripted memories during PE on day 2, the ketamine infusion procedure will begin inside the MRI. A physician will oversee and administer the ketamine infusions. A nurse will accompany the subject throughout the study sessions, from the insertion of bilateral cannula for drug infusion and blood sampling, to the recovery following ketamine infusion. Whilst subjects undergo the infusion, their heart rate and blood pressure will be constantly monitored. The participant will receive a steady state ketamine infusion of 0.50 mg/kg/hour. The infusion will continue for 40 minutes.
  Interventions: Drug: Ketamine
- Midazolam with prolonged exposure (Active Comparator): After the reactivation of the scripted memories during PE on day 2, the midazolam infusion procedure will begin inside the MRI. A physician will oversee and administer the Midazolam infusions. A nurse will accompany the subject throughout the study sessions, from the insertion of bilateral cannula for drug infusion and blood sampling, to the recovery following midazolam infusion. Whilst subjects undergo the infusion, their heart rate and blood pressure will be constantly monitored. The participant will receive a steady midazolam infusions at a rate 0.045 mg/kg for 40 minutes.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — Prolonged exposure therapy combined with a single infusion of 0.50 mg/kg/hour for 40 min on day 2.
  Other Names: Ketalar
  Arms: Single infusion of Ketamine with prolonged exposure
Drug: Midazolam — Prolonged exposure therapy combined with a single infusion of 0.045 mg/kg/hour for 40 min on day 2.
  Other Names: Versed
  Arms: Midazolam with prolonged exposure

SUMMARY:
The purpose of this study is to combine a single infusion of Ketamine with 7-days of trauma focus psychotherapy to relieve post traumatic stress disorder (PTSD) symptoms more effectively. This treatment has the potential to produce a significant therapeutic effect that otherwise would take months to occur.

DETAILED DESCRIPTION:
Based on the current research findings on the therapeutic effectiveness of trauma focus psychotherapy and of ketamine, combining the two treatments may yield a promising new rapid 7-day treatment for PTSD. As PTSD symptoms' structure is comprised of several unique clusters which include re-experiencing, avoidance, numbing/depression and hypervigilance the investigators hypothesize that by combining Ketamine with prolonged exposure (PE) the investigators can address these symptoms clusters more effectively. This treatment has the potential to produce a significant therapeutic effect that otherwise would take months to occur by tapping on the enhanced neuroplasticity and the antidepressant effect of ketamine (which lasts between 24hrs to 7 days), to promote rapid changes in learning and memory using prolonged exposure therapy within this unique "window of opportunity".

During the first visit participants will undergo a clinical interview to establish a PTSD diagnosis and other eligibility criteria. If found eligible participants will be invited to take part in this 7-day rapid treatment trial for PTSD.

On the first therapy visits, participants will be educated about the psychological treatment that will be provided and the potential benefit of ketamine to enhance the psychotherapy outcomes.

On the second day of the study, participants will receive an infusion of ketamine or placebo and will undergo a magnetic resonance imaging (MRI) scan and will receive the second psychotherapy session.

On days 3-6 participants will attend a 60-90 minutes psychotherapy session to address their PTSD symptoms.

Day 7 will include another MRI scan and the last psychotherapy session.

Participants will be asked to come back for a follow up evaluation of their PTSD symptoms 30 and 90 days post discharge.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 21-75 years. This age range was chosen to fit with prior samples in which no adverse effects of ketamine have been observed. Adults in the 18-20 ranges have been eliminated because previous experience indicates that they often lack the maturity to participate effectively in similar protocols. Females will be included if they are not pregnant and agreed to utilize a medically accepted birth control method (to include oral, injectable, or implant birth control, condom, diaphragm with spermicide, intrauterine device, tubal ligation, abstinence, or partner with vasectomy) or if post-menopausal for at least 1 year, or surgically sterile.
* Able to provide written informed consent according to Yale HIC guidelines.
* Able to read and write English as a primary language.
* Diagnosis of PTSD, as determined by the Clinician Administered PTSD Scale (CAPS-5) (Weathers et al., 2013).
* Must have a score of 50 or higher on the Clinician-Administered PTSD Scale (CAPS-5) at screening.
* No more than mild Traumatic Brain Injury (TBI) according to a modified version of the Brief TBI Screen (Schwab, et al., 2006).
* Must not have a medical/neurological problem or use medication that would render ketamine unsafe by history or medical evaluation.

Exclusion Criteria:

* Patients with a diagnostic history of bipolar disorder, schizophrenia or schizoaffective disorder or currently exhibiting psychotic features as determined by the Structured Clinical Interview for DSM (SCID) (First, et al. 2010); dementia or suspicion thereof, are excluded. Other DSM Axis I disorders are permitted as long as they are not considered primary disorders.
* Patients with a history of antidepressant-induced hypomania or mania as determined by open-ended psychiatric interview.
* Serious suicide or homicide risk, as assessed by evaluating clinician; A serious suicide risk will be considered an inability to control suicide attempts, imminent risk of suicide in the investigator's judgment, or a history of serious suicidal behavior, which is defined using the Columbia-Suicide Severity Rating Scale (C-SSRS) (Posner et al., 2011) as either (1) one or more actual suicide attempts in the 3 years before study entry with the lethality rated at 3 or higher, or (2) one or more interrupted suicide attempts with a potential lethality judged to result in serious injury or death.
* Substance abuse or dependence during the 6 months prior to screening as determined by the Structured Clinical Interview for DSM (SCID).
* Any significant history of serious medical or neurological illness.
* Any signs of major medical or neurological illness on examination or as a result of electrocardiogram (ECG) screening or laboratory studies.
* Lifetime history of psychoactive substance or alcohol dependence or substance or alcohol abuse (other than nicotine or caffeine abuse), or drinking more than 5 drinks/week during the last year.
* Abnormality on physical examination. A subject with a clinical abnormality may be included only if the study physician considers the abnormality will not introduce additional risk factors and will not interfere with the study procedure.
* A positive pre-study (screening) urine drug screen or, at the study physician's discretion on any drug screens given before the scans.
* Pregnant or lactating women or a positive urine pregnancy test for women of child-bearing potential at screening or prior to any imaging day.
* Positive HIV or Hepatitis B tests. This test will take place at the screening visit. Subjects will be invited back to the Yale Depression Research Program either for their next study visit or for a HIV/Hep debriefing session. A study physician will inform them in person of the results. They will be given access to counselling and advised of the appropriate next steps.
* Has received either prescribed or over-the-counter (OTC) centrally active medicine or herbal supplements within 60 days of enrollment into the study. Subjects who have taken OTC medication or herbal supplements may still be entered into the study, if, in the opinion of the principal/co-investigator, the medication received will not interfere with the study procedures or compromise safety.
* Any history indicating learning disability, mental retardation, or attention deficit disorder.
* Known sensitivity to ketamine.
* Body circumference of 52 inches or greater.
* Body weight of 250 pounds or greater.
* History of claustrophobia.
* Presence of cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies in vulnerable positions as assessed by a standard pre-MRI screening questionnaire.
* Donation of blood in excess of 500 mL within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-12; Primary Completion 2021-11-28 (Actual); Study Completion 2021-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Harpaz-Rotem, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Data from the initial stage of the investigation will be used to establish support for a Phase 3 RCT.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Infusion of Ketamine With Prolonged Exposure | Midazolam With Prolonged Exposure
Started | 14 | 14 (1 participant immediately withdrew after the first infusion session.)
End of Treatment (7 Days) | 13 | 13
30 Days Follow Up | 13 | 11
90 Days Follow Up | 11 | 10
Completed | 11 | 10
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Infusion of Ketamine With Prolonged Exposure | Midazolam With Prolonged Exposure | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (10.7) | 35.1 (10.3) | 38.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 1 | 2
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Symptoms
Description: PTSD symptoms severity will be evaluated overtime using the PTSD Checklist for DSM-5 (PCL-5), a 20 items self-report measure. Items are scored 0-4 (0=not at all to 4=Extremely), thus total PCL-5 score ranges from 0 to 80. Higher scores reflect greater severity of PTSD.
  Total PCL-5 scores are reported. PCL score>33 indicates probable PTSD diagnosis. Evidence for the PCL suggested 5 points reduction as a minimum threshold for determining whether an individual has responded to treatment and 10 points reduction in the PCL-5 as a minimum threshold for determining whether the improvement is clinically meaningful.
Time Frame: Baseline, 7 days, 30 days and 90 days
Population: The number that completed each assessment are presented and summarized- one participant in Midazolam arm was not included due to drop out prior to first assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Infusion of Ketamine With Prolonged Exposure | Midazolam With Prolonged Exposure
Number analyzed (Participants) | 14 | 13
score on a scale
  Baseline | 48.8 (12.3) | 44.4 (14.4)
  End of Treatment (7 days): number analyzed (Participants) | 13 | 13
  End of Treatment (7 days) | 29.5 (20.7) | 35.1 (16.8)
  30 Days Follow Up: number analyzed (Participants) | 13 | 11
  30 Days Follow Up | 32.7 (14.9) | 28.5 (17.2)
  90 Days Follow Up: number analyzed (Participants) | 11 | 10
  90 Days Follow Up | 34.2 (18.6) | 28.7 (18.3)

2. Secondary Outcome: Change in Beck Depression Inventory (BDI-II)
Description: The self-report BDI-II will be used to assess severity of depressive symptoms. A higher score is associated with higher severity of depression. The score is interpreted as follows: 0-13 indicates minimal depression, 14-19 indicates mild depression, 20-28 indicates moderate depression and 29-63 indicates severe depression
Time Frame: Baseline, 7 days, 30 days and 90 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Infusion of Ketamine With Prolonged Exposure | Midazolam With Prolonged Exposure
Number analyzed (Participants) | 14 | 13
score on a scale
  Baseline | 48.5 (5.7) | 47.6 (13.3)
  End of Treatment (7 Days): number analyzed (Participants) | 13 | 13
  End of Treatment (7 Days) | 38.9 (13.7) | 39.9 (11.8)
  30 Days Follow Up: number analyzed (Participants) | 13 | 11
  30 Days Follow Up | 43.0 (12.0) | 36.5 (12.0)
  90 Days Follow Up: number analyzed (Participants) | 11 | 10
  90 Days Follow Up | 42.8 (11.4) | 36.8 (15.8)

ADVERSE EVENTS:
Time Frame: Up to 90 days follow up.
Arm/Group | Single Infusion of Ketamine With Prolonged Exposure | Midazolam With Prolonged Exposure
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

LIMITATIONS AND CAVEATS:
Due to study termination, full enrollment was not achieved and therefore the intended regression modeling was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT02727998/Prot_SAP_000.pdf